CLINICAL TRIAL: NCT00526422
Title: Assessment of Caries Diagnosis & Caries Treatment
Brief Title: DPBRN Assessment of Caries Diagnosis & Caries Treatment
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: Kaiser Permanente (Other); Kaiser Foundation Hospitals, Center for Health Research (Other); University of Copenhagen (Other); University of Florida (Other); University of Alabama at Birmingham (Other); University of North Carolina (Other)
Other Study IDs: 101884
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Dental Caries
Keywords: Questionnaire, dental caries, diagnosis,treatment
MeSH Terms: conditions — Dental Caries; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Dental Preventive

SUMMARY:
The purpose of this study was to determine what methods Dental PBRN dentists use for diagnosis, prevention, and treatment of dental decay.

DETAILED DESCRIPTION:
The purpose of this project was to identify methods that Dental Practice-Based Research Network (DPBRN) dentist used to diagnose and treat caries lesions. The aims of the "Assessment of caries diagnosis and caries treatment" study were to: (1) quantify the percentages of DPBRN dentists who reported using selected methods for caries diagnosis; (2) quantify the percentage of DPBRN dentists who reported using a caries-risk assessment protocol of any variety; (3) quantify the percentages of DPBRN dentists who reported intervening surgically at carious states E1, E2, D1, D2, or D3; and (4) test the hypothesis that reported use of a caries-risk assessment protocol was associated with a higher likelihood of reporting use of a preventive program.

The aims were met by enrolling at least 200 DPBRN practitioner-investigators in the study, each of whom completed a 10-page questionnaire about caries diagnosis and treatment assessment. Findings from "Assessment of Caries diagnosis and caries treatment" study will be related to treatment that is actually delivered as determined in "Reasons for placing the first restoration on permanent tooth surfaces" study and "Reasons for replacement or repair of dental restorations" study. This group of three studies will lay a critical foundation for subsequent intervention studies designed to move the latest scientific advances about caries diagnosis and treatment into daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Practitioner investigators must have been enrolled in DPBRN and do at least some restorative dentistry in their practices.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The questionnaire was administered to all enrolled DPBRN dentist practitioner-investigators, defined as those who had comptled a DPBRN Enrollment Questionnaire who were 22 years or older and do at least some restorative dentistry in their practice.
Sampling Method: Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2006-02; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
A questionnaire was used to quantify the percentages of DPBRN practitioner-investigators who use selected methods for caries diagnosis and caries treatment. | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Gregg H Gilbert, DDS, MBA, Study Chair — University of Alabama at Birmingham; Valeria V. Gordan, DDS, MS, Principal Investigator — University of Florida

REFERENCES:
- See also: Related Info — http://DentalPBRN.org
- See also: Related Info — http://DPBRN.org